CLINICAL TRIAL: NCT07079176
Title: Etomidate Combined With Propofol Versus Propofol for Sedation in High-Altitude Patients During Gastroscopy: a Randomized Multicenter Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-6-20
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Gastrointestinal Endoscopy
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EP group (Experimental)
  Interventions: Drug: etomidate combined with propofol
- P group (Active Comparator)
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: etomidate combined with propofol — Patients initially received oxygen via nasal cannula at 5 L/min. All patients underwent routine noninvasive monitoring of blood pressure, ECG, and oxygen saturation. In the EP group, patients received 50 μg fentanyl, followed by a slow intravenous injection of a propofol-etomidate mixture (10 mL:20 mg etomidate + 10 mL:100 mg propofol) at 0.1-0.2 mL/kg. Supplemental doses of 0.05 mL/kg were administered as needed to maintain sedation throughout the procedure.
  Arms: EP group
Drug: propofol — Patients initially received oxygen via nasal cannula at 5 L/min. All underwent routine noninvasive monitoring of blood pressure, ECG, and oxygen saturation. In the P group, 50 μg fentanyl was administered, followed by a slow intravenous injection of propofol (1-2 mg/kg) after 3 minutes. Supplemental doses of 0.5 mg/kg were administered as needed to maintain sedation throughout the procedure.
  Arms: P group

SUMMARY:
One of the most common adverse events during sedated gastrointestinal endoscopy is hypoxemia, which can lead to serious consequences. When sedated gastrointestinal endoscopy is performed in high-altitude regions with thin air and lower atmospheric pressure, the risk of hypoxemia in patients significantly increases. Traditionally, propofol is the primary agent for sedation during gastrointestinal endoscopy, offering rapid onset and recovery. However, propofol has many side effects, the most important of which is inhibition of respiration and hypotension. Etomidate has less effect on respiration compared to propofol. But there are also adverse reactions of etomidate such as muscular tremor, nausea and vomiting. This study aims to explore whether the etomidate combined with propofol anesthesia method can reduce the risk of hypoxemia during sedated gastrointestinal endoscopy in high-altitude regions, compared to the traditional propofol anesthesia method .

ELIGIBILITY:
Inclusion Criteria:

Age: 18 ≤ years ≤ 70 Patients undergoing pain-free gastroscopy or treatment Endoscopy duration within 30 minutes Informed consent obtained from patient or family member

Exclusion Criteria:

Concomitant diagnosis of cardiac diseases (e.g., heart failure, angina, myocardial infarction, arrhythmia) Diagnosed pulmonary diseases Liver diseases Kidney diseases Intracranial hypertension ASA class III or higher Concomitant active upper respiratory tract infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 732 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
The risk of hypoxemia | during sedated gastrointestinal endoscopy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31278907/